CLINICAL TRIAL: NCT02225847
Title: Effect of Gardening on Brain Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Foliage Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201400425
Record Dates: First submitted 2014-08-20; First posted 2014-08-26 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Stress; Depression; Anxiety; Quality of Life
Keywords: Gardening; Therapeutic Horticulture; Functional Magnetic Resonance Imaging; Psychometric Assessment; Stress; Depression; Anxiety; Quality of Life; Wellness
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Gardening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Members of this group will continue with their daily life activities and will not receive gardening intervention. The control group will be given a set of psychometric assessments for health and quality of life evaluations and undergo a Functional Magnetic Resonance Imaging (fMRI) brain scan, followed by a second round of psychometric assessments and a fMRI brain scan administered seven to eight weeks after the initial baseline psychometric assessments and fMRI brain scan.
  Interventions: Procedure: Functional Magnetic Resonance Imaging (fMRI); Behavioral: psychometric assessments
- Gardening (Experimental): Members of this group will be given a set of psychometric assessments for health and quality of life evaluations and a Functional Magnetic Resonance Imaging (fMRI) brain scan prior to receiving the gardening activities intervention. The gardening intervention will consist of twice weekly group sessions lasting 60 minutes in duration that will take place in a greenhouse. The duration of the experimental intervention will be six weeks for a total of 12 individual gardening activity sessions. Following the completion of the gardening intervention, a second round of psychometric assessments and a fMRI brain scan will be administered seven to eight weeks after the initial baseline psychometric assessments and fMRI brain scan.
  Interventions: Other: Gardening; Procedure: Functional Magnetic Resonance Imaging (fMRI); Behavioral: psychometric assessments

INTERVENTIONS:
Other: Gardening — The intervention consists of twice weekly group sessions of gardening activities of 60 minutes in duration that will take place in a greenhouse. A total of 12 gardening sessions administered over a period of six weeks will include planting seeds, bulbs and tubers, transplanting seedlings, vegetative propagation and sight, smell, taste and touch sensory based activities.
  Arms: Gardening
Procedure: Functional Magnetic Resonance Imaging (fMRI) — Functional magnetic resonance imaging will be employed to assess whether engaging in gardening activities in a greenhouse does or does not alter the spatial patterns of brain network activation relative to changes that occur between the groups.
Behavioral: psychometric assessments — The following assessments will be used: The SF-36 Health Survey assessment instrument (Ware and Sherbourne 1992; Hays et al 1993), the Beck Depression Inventory 2nd edition (BDI-II) (Beck et al 1988), The State Trait Anxiety Inventory (STAI) instrument (Form Y) (Spielberger et al 1983), the Profile of Mood States 2nd edition short form for adults instrument (POMS2-AS), and the Perceived Stress Scale (PSS) (Cohen et al 1983) for changes that occur in between the groups.

SUMMARY:
The objective of the research is to test the hypothesis that participating in group-based gardening activities alters brain network activation and function, and that such change occurring in the brain forms the neurobiological basis for much of the nonphysical activity portion of the therapeutic benefits of gardening and horticultural therapy. Assessment of the effects of the gardening activities on the experimental population will take two approaches, the first being the use of functional Magnetic Resonance Imaging (fMRI) to assess the regions of the brain that may become activated as a consequence of experiencing the cumulative gardening activities and associated stimuli. The allied approach will employ widely used and well-established self-reported assessment instruments that will capture information about the health and well-being that will then provide a psychometrically-based before and after physical and health summary of the participants in the control group and those engaged in the gardening activities.

DETAILED DESCRIPTION:
The goal of this project is to better understand how interacting and working with plants in a group gardening activities program that takes place in a greenhouse effects patterns of brain activity and overall health and well-being. There has been essentially no assessment of the effects of gardening or engaging in gardening activities on brain activity using functional MRI (fMRI) approaches. This study will employ visual stimuli to assess the effects of the gardening activities treatment on Blood Oxygen Level Dependent (BOLD) responses as revealed by fMRI in study subjects in a comparison of responses before and after engaging in the gardening intervention program.

Specifically this study seeks to determine whether engaging in gardening activities taking place in a greenhouse can influence brain activity and function, and result in changes in overall quality of life status of subjects in a wellness population.

The total study population (N = 23) will consist of 11 healthy women in the control group, and 12 healthy women in the treatment group. There will be fMRI brain scans and psychometric pre- and post-intervention assessments administered to the study subjects. The fMRI and psychometric assessments will be administered within 10 days prior to the start of the intervention, and within 10 days following the completion of the treatment intervention. The control group will continue with normal daily life over a seven to eight week interval, and receive no other intervention. The treatment group will be divided into two groups of six women each that will receive the gardening intervention on different days of the week. The participants in the treatment group will receive an experimental intervention consisting of 12 gardening sessions, each approximately 60 minutes in duration over a six week treatment period. Each gardening session will take place at the same time of day twice each week, and follow a standardized programming sequence to ensure equivalency of intervention across all gardening sessions. Ambient environmental conditions in the greenhouse during the gardening sessions will be monitored and recorded. The gardening activities will emphasize growing plants from seeds, plant propagation techniques, transplanting, and plant-mediated taste, visual, olfactory and touch sensory stimulation. All gardening sessions will begin with a short educational module introducing the plants and gardening activities taking place during each session. In addition to the pre- and post-intervention assessments, psychometric assessments will be administered for depression and mood states at specific time points during the gardening activities to the treatment group to evaluate any changes over time resulting from the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* 26 - 49 years of age
* Not pregnant
* Non-gardener
* Non-smoker
* Good Health
* Able to participate in all aspects of the study, including working with plants.

Exclusion Criteria:

* Uncomfortable in close spaces (claustrophobia)
* Allergies to plants
* Allergies to plant parts like pollen
* Allergies to plant-based foods
* No additions to alcohol or to recreational drugs or prescription medications
* Not suffering from recurring pain, and
* No diseases, disorders or disabilities that affect daily life.

Ages: 26 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in Spatial Patterns of Brain Network Activation | Baseline, up to 2 months
  Functional magnetic resonance imaging will be employed to assess whether engaging in gardening activities in a greenhouse does or does not alter the spatial patterns of brain network activation relative to changes that occur in the control group.

SECONDARY OUTCOMES:
Change in Overall Health Status | Baseline, up to 2 months
  The SF-36 Health Survey assessment instrument (Ware and Sherbourne 1992; Hays et al 1993) will be used to evaluate eight scales that link to physical and mental health over a 4-week recall interval. This will reveal whether engaging in gardening activities will or will not result in changes in the overall health status based on instrument's physical and mental health subcomponent assessments of the gardening treatment group compared to the control group. The overall assessment scale for the SF-36 ranges from a low of 36 to a high of 400, with the U.S. norm being 314.
Change in Depressive Symptomatology | Baseline, up to 2 months
  The study protocol will use the Beck Depression Inventory 2nd edition (BDI-II) (Beck et al 1988) with a recall interval of 2-weeks to gain insight relative to the intensity of depression. This assessment will determine whether engaging in gardening will or will not result in changes in depressive symptomatology of the gardening treatment group relative to the control group. The assessment scale for the Beck BDI ranges from a low of 10 to a high of 63. Scores 0-13 indicate minimal depressive symptomatology and above 19 up to 63 moderate to severe depressive symptomatology.
Change in State Anxiety | Baseline up to 2 months
  The State Trait Anxiety Inventory (STAI) instrument (Form Y) (Spielberger et al 1983) will be used in this study to gain insight regarding the relative intensity of anxiety being experienced by the gardening treatment group relative to the control group. The STAI reports on "at this moment" status. The STAI assessment will seek to determine whether engaging in gardening will or will not result in changes in State Anxiety status of the participants. The overall assessment scale for the STAI-Y ranges from a low of 20 to a high of 80, with higher scores indicating greater intensity of anxiety.
Change in Mood States | Baseline, up to 2 months
  The study protocol will employ the Profile of Mood States 2nd edition short form for adults instrument (POMS2-AS) with an immediate recall interval (McNair et al 1981; Shacham 1983) to gain insight of the relative to transient and fluctuating moods and enduring states of affect. The POMS2-AS will assess whether engaging in gardening activities will or will not result in changes in mood and enduring states of affect status of the gardening treatment group relative to the control group, both during and following the completion of the gardening activities treatment regimen. The assessment scale for the POMS2-AS ranges from 5 to a high of 100 per scale .
Change in Perceived Stress | Baseline, up to 2 months
  The study will use the Perceived Stress Scale (PSS) (Cohen et al 1983) with a recall interval of 4-weeks to gain insight relative to the intensity of perceived stress. This assessment will determine whether engaging in gardening activities will or will not result in changes in the perceived stress levels of the gardening treatment group relative to the control group. The assessment scale for the Perceived Stress Scale ranges from a low of 0 to a high of 40, indicating higher stress at higher scores. The norm score for women is 13.7.

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Guy, PhD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - Fifield Hall, Gainesville, Florida
  - McKnight Brain Institute, Gainesville, Florida
  - Wilmot Greenhouse, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Yes
At the completion of the study de-identified raw fMRI data from the study will be submitted to OpenfMRI, an open source fMRI database repository located at: https://openfmri.org/.
  De-identified processed datasets from the brain scans will be submitted to BrainMap or Neurosynth for open source access suitable for meta-analysis of processed fMRI data from brain imaging studies. The URL for BrainMap: http://www.brainmap.org/.
  The URL for Neurosynth is: http://www.neurosynth.org/.

REFERENCES:
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Beck, AT, Steer RA, Garbin MG. Psychometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clinical Psychology Review 1988 (8):77-100.
- [Background] Spielberger, CD, Gorsuch RL, Lushene R. The State-Trait Personality Inventory STAI-Y, form Y. Consulting Psychologists Press, Palo Alto. 1983
- [Background] McNair PM, Lorr M, Droppleman LF. POMS manual (2nd ed.). San Diego: Educational and Industrial Testing Service. 1981.
- [Background] Shacham S. A shortened version of the Profile of Mood States. J Pers Assess. 1983 Jun;47(3):305-6. doi: 10.1207/s15327752jpa4703_14. PMID 6886962
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417